CLINICAL TRIAL: NCT07231887
Title: Effect of Different Positions During Extubation on Incidence of Hypoxemia in the Peri Extubation Period of Pediatric OSAS Surgery Under General Anesthesia, Randomized Controlled Trial
Brief Title: Effect of Different Positions During Extubation on Incidence of Hypoxemia in the Peri Extubation Period
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Abbas Hassan, Ass. Prof., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ENT2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (lateral position): (Active Comparator): ENT surgery patients positioned laterally with head in zero position after completion of surgery and before extubation till full recovery and discharge from PACU.
  Interventions: Procedure: positioning during peri-extubation
- Group S (Sim' position): (Active Comparator): ENT surgery patients positioned in semi-prone position after completion of surgery and before extubation till full recovery and discharge from PACU.
  Interventions: Procedure: positioning during peri-extubation

INTERVENTIONS:
Procedure: positioning during peri-extubation — investigate and compare whether the use of lateral position or semi-prone position impact on the occurrence of choking, agitation, decreased pulse oxygen saturation - (SpO2) and the oral and nasal secretions during the awakening period.

SUMMARY:
Pediatric Obstructive Sleep Apnea Syndrome (OSAS) is common, often due to enlarged tonsils/adenoids. Tonsillectomy/adenoidectomy frequently performed under GA with tracheal intubation due to the age of children. Risk of hypoxemia and respiratory complications during the peri-extubation period is high.

DETAILED DESCRIPTION:
The most common disorder of sleep apnea in children is obstructive sleep apnea syndrome (OSAS), characterized by interrupted breathing and partial or complete obstruction of the upper airway, the main factor is the enlargement of the tonsils and adenoids in the pediatric pharynx. The clinical symptoms are snoring, and open-mouth breathing, then resulting in hypoventilation and hypoxemia. Due to the age of children, tonsillectomy and adenoidectomy are often performed under general anesthesia with tracheal intubation. The risk of hypoxemia and the degree of oxygen saturation reduction are bigger when the mask was removed in the supine position, and the most serious complication also occurred in the supine position. Therefore, the lateral position is preferable to the supine position for mask removal. There are few reports on the effect of different positions on complications related to tracheal extubation after tonsillectomy and adenoidectomy under general anesthesia in children with OSAS. In this study, we will investigate and compare whether the use of lateral position or semi-prone position impact on the occurrence of choking, agitation, decreased pulse oxygen saturation - (SpO2) and the oral and nasal secretions during the awakening period.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-10 years
* American Society of Anesthesiologists physical status classification (ASA) I - II
* Patients scheduled for ENT procedures involving tonsillectomy, adenoidectomy or adenotonsillectomy

Exclusion Criteria:

* • Patient legal guardian refusal to participate in the study.

  * Children with cardio-pulmonary disease

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 262 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxemic events in the peri-extubation period | one hour after extubation
  Hypoxemic events which last > 2 seconds after extubation will be recorded when Spo2 is less than 94% on room air.

SECONDARY OUTCOMES:
Incidence of respiratory complications | one hour after extubation
  Incidence of respiratory complications such as choking, laryngospasm, posterior tongue drop.

CONTACTS AND LOCATIONS:
Overall Officials: Shimaa A. Abbas, M.D., Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No